CLINICAL TRIAL: NCT04854278
Title: Development of Strategies to Identify, Analyse and Prevent Errors in the Vascular Hybrid Room - an Inter-professional Approach to Enhance Technical and Non-technical Performance and to Improve Patient Safety
Brief Title: Introduction of an Operating Room Black Box to Identify, Analyse and Prevent Errors in the Vascular Hybrid Room
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: BC-02220
Record Dates: First submitted 2021-04-02; First posted 2021-04-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Patient Safety; Endovascular Procedures; Quality Improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pilot study: Pilot study with 22 cases, no intervention
- Baseline measurement: Baseline measurement of +/- 100 cases, no intervention
- Post measurement: Post measurement of +/- 100 cases after implementation of a Massive Open Online Course
  Interventions: Other: Massive Open Online Course (MOOC)
- Registry of endovascular cases: Starting 1 january 2023

INTERVENTIONS:
Other: Massive Open Online Course (MOOC) — Combination of knowledge training with video scenarios and game-based learning provided to endovascular team members: surgeons, nurses and anesthetists
  Other Names: Radiation Safety in the hybrid room: the do's and don'ts
  Groups: Post measurement

SUMMARY:
The "OR Black box", an inclusive multiport data capturing system has been developed and successfully used for detailed analysis of laparoscopic surgical procedures. A pilot study has shown that this system can be successfully installed in the hybrid room at Ghent University Hospital and used for detailed analysis of intra-operative errors and radiation safety issues in endovascular procedures.

Secondary analysis of pilot study data via direct video coding assessed the relationship between leadership style of the surgeon and team behavior and possible fluctuations during surgery.

This novel approach allows a prospective objective assessment of human and environmental factors as well as measurement of errors, events and outcomes. In this study, the aim is to use the acquired knowledge to characterize a chain of events, identify high-risk interventions and identify areas for improvement, both on an organizational, team or individual level.

Hypothesis: non-technical skills, environmental factors and teamwork in the hybrid room correlate with surgical technical performance and error rates. Furthermore, we hypothesize that incidents and adverse events can be tracked to a chain of errors that is influenced by technical and non-technical skills as well as environmental factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective (planned more than 48 hours) endovascular procedures.
* Symptomatic aortic-iliac-femoral-popliteal-below the knee atherosclerotic stenotic or occlusive disease (PVI)
* Endovascular exclusion of thoracic aortic, infrarenal abdominal aortic and/or iliac aneurysm repair (EVAR)

Exclusion Criteria:

* No consent of patient
* No consent of all endovascular team members
* Emergency procedure (planned < 48h before)
* Endovascular procedure not treating atherosclerotic aortic-iliac-femoral-popliteal-below the knee disease or aortic-iliac aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for endovascular intervention at Ghent University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Error | Intraoperative errors will be measured per case through study completion, an average of 1.5 years.
  Evaluate errors during elective endovascular procedures in a hybrid room (error rate)

SECONDARY OUTCOMES:
Technical skills - PVI | Through study completion, an average of 1.5 years
  Assess technical skills of the surgeon on Global rating scale (range: 8-40) (the higher the score, the better)
Technical skills - EVAR - GRS | Through study completion, an average of 1.5 years
  Assess technical skills of the surgeon on Global rating scale (GRS) (range: 8-40) (the higher the score, the better)
Technical skills - EVAR - PRS | Through study completion, an average of 1.5 years
  Assess technical skills of the surgeon on Procedure Specific rating scale (PRS) (range: 7-35) (the higher the score, the better)
Technical skills - EVAR - EVARATE | Through study completion, an average of 1.5 years
  Assess technical skills of the surgeon on EVARATE (EndoVascular Aortic Repair Assessment of Technical Expertise) (range: 7-35) (the higher the score, the better)
Non-technical skills - surgical team | Through study completion, an average of 1.5 years
  Assess non-technical skills of the surgeon via NOTSS (Non-Technical Skills for Surgeons)
Non-technical skills - nursing team | Through study completion, an average of 1.5 years
  Assess non-technical skills of the surgeon via SPLINTS (Non-technical skills of the scrub practitioner)
Distractions - auditory | Through study completion, an average of 1.5 years
  Assess distractions in the hybrid room: DiSI (Distractions in surgery index). Number and type of Auditory distractions
Distractions - people | Through study completion, an average of 1.5 years
  Assess distractions in the hybrid room: DiSI (Distractions in surgery index). Maximal number of people in the room
Distractions - doors | Through study completion, an average of 1.5 years
  Assess distractions in the hybrid room: DiSI (Distractions in surgery index). Number of times doors open
Radiation Safety - dose DAP | Through study completion, an average of 1.5 years
  Assess radiation safety dose: Dose Area Product (DAP)
Radiation Safety - dose AK | Through study completion, an average of 1.5 years
  Assess radiation safety dose: Air Kerma (AK)
Radiation Safety - fluoroscopy time | Through study completion, an average of 1.5 years
  Assess radiation safety dose: Fluoroscopy time (FT)
Radiation Safety - behavior | Through study completion, an average of 1.5 years
  Assess radiation safety behavior: Radiation safety scale (Range: 11-55) (the higher the score, the better)
Error work culture | Through study completion, an average of 1.5 years
  Assess error work culture in the hybrid room via a baseline survey: 10 items, each scored on a 5-Point Likert scale
Psycho-social well-being | Through study completion, an average of 1.5 years
  Assess psycho-social well-being of teammembers in the hybrid room via a pre and post procedure survey for each case
Incident reports | Through study completion, an average of 1.5 years
  Assess number of incident reports (obligatory existing platform in the hospital to report incidents) during Operation Black Black Box (ORBB) cases - incident rate
Technical Readiness and Acceptance | january 2023 until december 2025
  Team's technical readiness and acceptance towards a new technology (Lumiguide) in the hybrid operating room
Cognitive load | From January 1st 2023 until January 1st 2025
  Measured using the NASA-TLX

OTHER OUTCOMES:
Team behavior | Through study completion, an average of 1.5 years
  Assessment of team behavior indicators (speaking up, knowledge sharing, collaboration) via direct video coding
Leadership style | Through study completion, an average of 1.5 years
  Assessment of leadership style according to the 'full range of leadership' theory via direct video coding

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gordon L, Soenens G, Doyen B, Sunavsky J, Wheatcroft M, de Mestral C, Palter V, Grantcharov T, Van Herzeele I. Step, Error, and Event Frameworks in Endovascular Aortic Repair. J Endovasc Ther. 2022 Dec;29(6):937-947. doi: 10.1177/15266028211068768. Epub 2022 Jan 11. PMID 35012393
- [Result] Soenens G, Marchand B, Doyen B, Grantcharov T, Van Herzeele I, Vlerick P. Surgeons' Leadership Style and Team Behavior in the Hybrid Operating Room: Prospective Cohort Study. Ann Surg. 2023 Jul 1;278(1):e5-e12. doi: 10.1097/SLA.0000000000005645. Epub 2022 Jul 29. PMID 35904023
- [Result] Soenens G, Doyen B, Vlerick P, Hertault A, Maurel B, Kellens PJ, Bacher K, Van Herzeele I; VESTA (Vascular surgery in Europe radiation SafeTy Alliance). Development, Feasibility, and Knowledge Impact of a Massive Open Online Course on Radiation Safety: A Multicentre Prospective Cohort Study. Eur J Vasc Endovasc Surg. 2024 May;67(5):838-846. doi: 10.1016/j.ejvs.2023.11.047. Epub 2023 Dec 1. PMID 38042252
- [Result] Soenens G, Gorden L, Doyen B, Wheatcroft M, de Mestral C, Palter V, Van Herzeele I; ENDORATE-PVI consortium. Editor's Choice - Development and Testing of Step, Error, and Event Frameworks to Evaluate Technical Performance in Peripheral Endovascular Interventions. Eur J Vasc Endovasc Surg. 2024 Aug;68(2):227-235. doi: 10.1016/j.ejvs.2024.03.007. Epub 2024 Mar 15. PMID 38492630
- [Result] Soenens G, Vlerick P, Bacher K, Rennie N, Grantcharov T, Van Herzeele I. Impact of a Massive Open Online Course on Radiation Safety in the Hybrid Operating Room. Eur J Vasc Endovasc Surg. 2025 Nov;70(5):693-694. doi: 10.1016/j.ejvs.2025.07.002. Epub 2025 Jul 7. No abstract available. PMID 40633718
- [Result] Kaya J, Bonte E, Rennie N, Soenens G, Moreels N, Vlerick P, Van Herzeele I. Mapping Distractions in the Hybrid Operating Room During Elective Endovascular Aortic Procedures. World J Surg. 2025 Jun;49(6):1676-1682. doi: 10.1002/wjs.12605. Epub 2025 Apr 29. PMID 40302105
- [Result] Soenens G, Doyen B, Vlerick P, Vermassen F, Grantcharov T, Van Herzeele I. Assessment of Endovascular Team Performances Using a Comprehensive Data Capture Platform in the Hybrid Room: A Pilot Study. Eur J Vasc Endovasc Surg. 2021 Jun;61(6):1028-1029. doi: 10.1016/j.ejvs.2021.02.021. Epub 2021 Mar 17. No abstract available. PMID 33744093
- [Result] Doyen B, Gordon L, Soenens G, Bacher K, Vlerick P, Vermassen F, Grantcharov T, Van Herzeele I. Introduction of a surgical Black Box system in a hybrid angiosuite: Challenges and opportunities. Phys Med. 2020 Aug;76:77-84. doi: 10.1016/j.ejmp.2020.06.013. Epub 2020 Jun 29. PMID 32615511
- [Result] Doyen B, Soenens G, Maurel B, Hertault A, Gordon L, Vlerick P, Vermassen F, Grantcharov T, van Herzeele I. Assessing endovascular team performances in a hybrid room using the Black Box system: a prospective cohort study. J Cardiovasc Surg (Torino). 2023 Feb;64(1):82-92. doi: 10.23736/S0021-9509.22.12226-3. Epub 2022 Sep 28. PMID 36168949